CLINICAL TRIAL: NCT02522286
Title: Creating a Zone of Openness to Increase Patient-Centered Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Collaborators: Gordon and Betty Moore Foundation (Other); Dartmouth College (Other); University of Rochester (Other); Ideo (Industry); PRN Consulting (Unknown)
Responsible Party: Principal Investigator, Ming Tai-Seale, Phd, MPH, Senior Scientist, Palo Alto Medical Foundation
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 37930708; PCORI-1IP2PI000055-01 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2015-05-16; First posted 2015-08-13 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2017-09

CONDITIONS: Patient Engagement; Physician's Role; Physician-Patient Relationship
Keywords: patient engagement; physician's role; patient- centered care; communication
MeSH Terms: conditions — Patient Participation; Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual Care (No Intervention): Standard clinical care in primary care offices
- Ask 3 Questions (Experimental): Patients using 3 questions to their physicians when making medical decisions during the office visit.
  Interventions: Behavioral: Ask 3 Questions
- Open Communication (Experimental): This arm has three components: (1) Patients, physicians, and medical assistants watching a video aimed at encouraging open communication; (2) Patients fill out a Visit Companion Booklet about what are the most important issues they want to discuss with their physicians, record their next steps, and teach back on their next steps; (3) physicians receiving communication coaching from a Standardized Patient Instructor on patient-centered communication.
  Interventions: Behavioral: Open Communication
- Ask 3 Questions + Open Communication (Experimental): A combination of both the Ask 3 and Open Communication arms.
  Interventions: Behavioral: Ask 3 Questions; Behavioral: Open Communication

INTERVENTIONS:
Behavioral: Ask 3 Questions — Participants were asked to bring an "Ask 3" questions flyer into their appointment to use if they needed to make a choice about their health care during their appointment. These 3 questions have been shown to help patients make more informed decisions about their healthcare.
  Arms: Ask 3 Questions; Ask 3 Questions + Open Communication
Behavioral: Open Communication — Open Communication includes a combination of interventions. 1) Participants used a Visit Companion Booklet to write out issues they would like to discuss with their physician during their appointment before showing up. They were also asked to write out any next steps decided on during their appointment and to repeat back to their doctor what they wrote before leaving.
  2) Patients watched a short, informational cartoon video to better understand the Visit Companion Booklet.
  3) Participating physicians received a training through the use of a Standardized Patient Instructor as a means of providing convenient, individualized training on communication techniques. Dyads (physicians and their medical assistants) were trained on how to incorporate the Visit Companion Booklet into workflow.
  Arms: Ask 3 Questions + Open Communication; Open Communication

SUMMARY:
This study implements a simple evidence-based patient activation intervention - "Ask 3 Questions"- augmented by a novel theory-based intervention - "Open Communication" - aimed at activating patients and healthcare providers. The goal of this project is to increase patient and physician's preparedness for more having more questions, expressing differing opinions, and working collaboratively in making medical decisions that are both informed and responsive to patients' needs and preferences.

DETAILED DESCRIPTION:
Conduct a pilot randomized controlled trial (RCT) to compare two interventions, "Ask 3 Questions," "Open Communication," a combination of both "Ask 3 Questions" and "Open Communication," to a usual care control condition. These data will inform a potential future large scale evaluation of the interventions in clinical practice. Consistent with a patient-centered approach, outcome measures are selected in collaboration with a group of patient stakeholders and will include measures of patient satisfaction. The study aims to collect 75 post-visit surveys and 10 appointment audio-recordings from patients at each of 4 participating sites (a total of 300 post-visit surveys and 40 audio-recordings).

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a scheduled appointment with the participating family medicine and internal medicine physicians during the study period.

Exclusion Criteria:

* Non-English speakers
* Patients younger than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Tai-Seale, PhD, MPH, Principal Investigator — Palo Alto Medical Foundation

REFERENCES:
- [Background] Barr PJ, Thompson R, Walsh T, Grande SW, Ozanne EM, Elwyn G. The psychometric properties of CollaboRATE: a fast and frugal patient-reported measure of the shared decision-making process. J Med Internet Res. 2014 Jan 3;16(1):e2. doi: 10.2196/jmir.3085. PMID 24389354
- [Background] Lerman CE, Brody DS, Caputo GC, Smith DG, Lazaro CG, Wolfson HG. Patients' Perceived Involvement in Care Scale: relationship to attitudes about illness and medical care. J Gen Intern Med. 1990 Jan-Feb;5(1):29-33. doi: 10.1007/BF02602306. PMID 2299426
- [Background] Elwyn G, Hutchings H, Edwards A, Rapport F, Wensing M, Cheung WY, Grol R. The OPTION scale: measuring the extent that clinicians involve patients in decision-making tasks. Health Expect. 2005 Mar;8(1):34-42. doi: 10.1111/j.1369-7625.2004.00311.x. PMID 15713169
- [Result] Tai-Seale M, Elwyn G, Wilson CJ, Stults C, Dillon EC, Li M, Chuang J, Meehan A, Frosch DL. Enhancing Shared Decision Making Through Carefully Designed Interventions That Target Patient And Provider Behavior. Health Aff (Millwood). 2016 Apr;35(4):605-12. doi: 10.1377/hlthaff.2015.1398. PMID 27044959
- See also: Open Communication Video — http://link.brightcove.com/services/player/bcpid1275282370001?bckey=AQ~~,AAABC-FjqSk~,kZ8F7j6A7AFwKgMjgryyU9fin2L2jWOx&bctid=2952214672001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2014 to April 2015, 75 patients were screened and enrolled for each of the 4 participating family or internal medicine clinics. Researchers met with interested patients who had a regularly scheduled appointment in order to consent and advise on how to use the study materials. After their visit, they completed a post-visit survey.
Pre-assignment Details: New patients and patients with physical exams or osteopathic evaluations were initially excluded though later allowed for recruitment for some physicians at one of the participating clinics. There were 6 patients who consented to participate but did not complete the final survey when exiting their appointment.
Period: Overall Study
Arm/Group | Usual Care | Ask 3 Questions | Open Communication | Ask 3 Questions + Open Communication
Started | 78 | 75 | 75 | 78
Completed | 75 | 75 | 75 | 75
Not Completed | 3 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The number of participants that filled in the survey that was provided to them by researchers after their primary care provider appointment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Ask 3 Questions | Open Communication | Ask 3 Questions + Open Communication | Total
Number analyzed (Participants) | 75 | 75 | 75 | 75 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (16.2) | 50.7 (15.6) | 49.0 (15.0) | 61.4 (15.3) | 54.0 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 34 | 44 | 54 | 182
  Male | 25 | 41 | 31 | 21 | 118
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 45 | 38 | 44 | 63 | 190
  Asian or Pacific Islander | 15 | 24 | 20 | 3 | 62
  Other | 15 | 13 | 11 | 9 | 48

OUTCOME MEASURES:

1. Primary Outcome: Patient Rating of Shared Decision Making
Description: Responses from CollaboRATE, a 3-question validated patient reported measure of shared decision making. Patients answered questions on a scale of 0 ("definitely disagree") to 9 ("definitely agree"). The CollaboRATE questions are as follows: 1) How much effort was made to help you understand your health issues? 2) How much effort was made to listen to the things that matter most to you about your health issues?, 3) How much effort was made to include what matters most to you in choosing what to do next? The outcome measure was the percent of patients who gave the top score of 9 on all three questions.
Time Frame: Day 1 (outcomes measures were assessed once for each participant)
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Usual Care | Ask 3 Questions | Open Communication | Ask 3 Questions + Open Communication
Number analyzed (Participants) | 75 | 75 | 75 | 75
percentage of participants | 66.7 (17.0) | 72.0 (17.3) | 74.7 (14.0) | 74.7 (12.5)

2. Primary Outcome: Doctor Facilitation Subscale of the Perceived Involvement in Care Scale
Description: "Responses from this patient reported measure regarding their attitudes of doctor facilitation of patient involvement for their illness management. Patients rated 5 statements on a scale of 0 (""definitely disagree"") to 9 (""definitely agree""). The statements are as follows: 1) My doctor encouraged me to talk about personal concerns related to my medical symptoms, 2) My doctor asked me what I believe is causing my medical symptoms, 3) My doctor gave me a complete explanation for my medical symptoms or treatment, 4) My doctor encouraged me to give my opinion about my medical treatment, 5) My doctor asked me whether I agree with his/her decisions. The outcome measure was the percent of patients who gave the top score of 9 on all five statements.
Time Frame: Day 1 (outcomes measures were assessed once for each participant)
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Usual Care | Ask 3 Questions | Open Communication | Ask 3 Questions + Open Communication
Number analyzed (Participants) | 75 | 75 | 75 | 75
percentage of participants | 37.3 (16.6) | 42.7 (11.5) | 45.3 (12.7) | 46.7 (14.8)

3. Primary Outcome: Patient Responses to Stakeholder Generated Questions
Description: Patient responses to statements that were generated by the study's patient and physicians stakeholders regarding how they felt during their appointment. Patients rated 5 statements, described below, on a scale of 0 (definitely disagree) to 9 (definitely agree). The outcome measure is the percent of patients that responded with a top score of "9." Statement 1: My doctor and I accomplished my most important goals today. Statement 2: I feel cared for. Statement 3: I feel comfortable being open with my doctor. Statement 4: I felt my doctor was open with me. Statement 5: I know what my next steps are.
Time Frame: Day 1 (outcomes measures were assessed once for each participant)
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Usual Care | Ask 3 Questions | Open Communication | Ask 3 Questions + Open Communication
Number analyzed (Participants) | 75 | 75 | 75 | 75
percentage of participants
  Statement 1 (n=75) | 86.7 (12.6) | 96.0 (6.3) | 90.5 (11.4) | 81.3 (10.3)
  Statement 2 (n=75) | 81.3 (10.4) | 93.2 (8.2) | 89.2 (11.5) | 81.1 (11.6)
  Statement 3 (n=75) | 80.0 (9.2) | 96.0 (6.0) | 90.7 (9.4) | 83.6 (12.6)
  Statement 4 (n=75) | 83.8 (7.7) | 90.5 (10.1) | 92.0 (9.1) | 85.3 (11.7)
  Statement 5 (n=75) | 82.2 (11.7) | 87.7 (7.8) | 91.8 (8.6) | 81.9 (12.5)

4. Primary Outcome: Patients' Feeling of Respect by Their Doctor
Description: Patient responses to one statement modified from Consumer Assessment of Healthcare Providers and Systems (CAHPS) regarding the respect they felt from their doctor. Patients rated the statement "My doctor showed respect for what I had to say," on a scale of 1 ("definitely disagree") to 4 ("definitely agree"). The outcome measure was the percentage of patients that gave the top score of 4 on this statement.
Time Frame: Day 1 (outcomes measures were assessed once for each participant)
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Usual Care | Ask 3 Questions | Open Communication | Ask 3 Questions + Open Communication
Number analyzed (Participants) | 75 | 75 | 75 | 75
percentage of participants | 96.0 (4.6) | 98.7 (3.0) | 97.3 (2.4) | 90.7 (6.6)

5. Secondary Outcome: Option 5 Shared Decision Making Score
Description: Researchers measured the shared decision making process that occurs between patients and physicians during the appointment using a method called OPTION5. Researchers listened to audio-recorded patient appointments, identified any topic, defined as "a health issue where alternate treatment or management option exist/where the need for a decision exists," and then measured each topic for each of the OPTION5 items on a scale of 0 ("no effort: nothing observed or heard") to 20 (exemplary effort: excellent, careful attention to communication around the ideas and issues, with checks on understanding," for each of the 5 items described below. The total score is a sum of the scores from each of the 5 items at the clinic.
  Item 1: presenting options Item 2: establishing a partnership with the patient Item 3: describing pros and cons of options Item 4: eliciting patient preferences Item 5: integrating patient preferences into the decision
Time Frame: Day 1 (outcomes measures were assessed once for each participant based on analysis of the audio recording of their visits)
Population: From the 75 patients at each of the 4 clinics, 10 appointments were randomly selected to be audio-recordinged. The Number of Participants Analyzed reflects the number of topics identified from the 10 recordings at each clinic.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | Ask 3 Questions | Open Communication | Ask 3 Questions + Open Communication
Number analyzed (Participants) | 51 | 49 | 48 | 52
scores on a scale
  Item 1 (out of 20) | 6.7 (2.6) | 7.7 (3.2) | 7.6 (2.9) | 6.4 (2.6)
  Item 2 (out of 20) | 4.1 (3.0) | 4.9 (3.5) | 4.9 (3.8) | 3.3 (3.1)
  Item 3 (out of 20) | 5.6 (3.6) | 7.2 (4.3) | 6.7 (4.3) | 5.8 (3.8)
  Item 4 (out of 20) | 3.8 (3.2) | 4.5 (3.8) | 5.1 (3.8) | 4.6 (4.0)
  Item 5 (out of 20) | 3.7 (3.2) | 4.4 (3.7) | 5.0 (3.8) | 4.4 (3.8)
  Overall Score (out of 100) | 23.9 (11.8) | 28.8 (16.8) | 29.2 (16.8) | 24.5 (14.6)

ADVERSE EVENTS:
Arm/Group | Usual Care | Ask 3 Questions | Open Communication | Ask 3 Questions + Open Communication
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75 | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75 | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No